CLINICAL TRIAL: NCT04861363
Title: Follow up of Ticagrelor Treatment Patterns in Chinese Acute Coronary Syndromes Patients- A Database Retrospective Study
Brief Title: Follow up of Ticagrelor Treatment Patterns in Chinese Acute Coronary Syndromes Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Yong Huo, Former director of the Department of cardiology, Principal Investigator, Clinical professor, Peking University First Hospital
Other Study IDs: ESR-18-13975
Record Dates: First submitted 2021-04-10; First posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a retrospective, observational, descriptive study which will include patients hospitalized for acute coronary syndrome (ACS) and treated with ticagrelor at discharge. Participants will come from the follow-up program of ACS patients taking ticagrelor 90 mg twice a day as part of the dual antiplatelet therapy at discharge. The primary objectives were to describe the ticagrelor treatment patterns-Ticagrelor persistence, discontinuation, switching, interruption and reasons in Chinese ACS patients; and also to describe 1-year clinical outcomes (Composite of any cause death, myocardial infarction, and stroke) of Chinese ACS patients in real-life practice based on ACS patient follow-up program database.

DETAILED DESCRIPTION:
Background： There are at least 2.5 million acute coronary syndromes (ACS) patients in China per year. Limited data about long term ticagrelor treatment patterns and clinical outcomes in Chinese ACS patients due to the lack of large high quality follow up database. This study is based on real-life practice and ticagrelor is prescribed according to the Chinese guideline and it takes place in real life.

Objective of this study:

Primary Objectives:

1. To describe the ticagrelor treatment patterns-Ticagrelor persistence, discontinuation, switching, interruption and reasons for discontinuation/switching/interruption in Chinese ACS patients.
2. To describe 1-year clinical outcomes (Composite of any cause death, myocardial infarction, and stroke) of Chinese ACS patients in real-life practice based on ACS patient follow-up program database.

Secondary Objectives:

1. To describe the impact of ticagrelor treatment pattern on clinical outcomes. (No confirmed conclusions regarding the efficacy or impact of ticagrelor treatment patterns will be drawn because of descriptive analysis.)
2. To analyze influence factors (age, region, hypertension, diabetes, chronic kidney disease (CKD), smoking, education, insurance etc) related to clinical outcomes

Exploratory Objectives:

To explore the influence factors (age, region, education, insurance, event, etc.) with ticagrelor treatment pattern; Analysis of other possible factors (such as smoke, low density lipoprotein-chlesterol [LDL-C]) affecting the prognosis of patients with ACS; Analysis of possible interactions and their influences between different factors associated with the prognosis of patients with ACS

Study design:

This is a retrospective, observational, descriptive study which will include patients hospitalized for ACS and treated with ticagrelor at discharge.

Data source：

Study participants： Participants will come from the follow-up program of ACS patients taking ticagrelor 90 mg twice a day as part of the dual antiplatelet therapy at discharge. During the follow-up period for 12 months after discharge. Telephone follow-up will be done 1, 3, 6, 12 months after discharge according to a structured questionnaire assessing the primary and secondary objectives of this study. Telephone interviews will be performed by the local ACS patient follow-up program assistants (nurses who enters information in the websites).

Study Variables:

Primary variables:

1. Ticagrelor treatment patterns-Ticagrelor persistence, discontinuation, switch, interruption and reasons for switching/discontinuation/interruption

1. Ticagrelor persistence: Proportion of patients who is on ticagrelor treatment every month after discharge; Duration of time from initiation to discontinuation of therapy.
2. Proportion of patients with ticagrelor discontinuation, switching and interruption and related reasons; Discontinuation of medications was defined as a break for P2Y12 at least three months; Switching means from Ticagrelor/Clopidogrel to another P2Y12 inhibitor (Clopidogrel to ticagrelor means re-switching if they were recorded). Interruption was defined as Ticagrelor discontinuation for more than 1 day and less than 3 months) 2. Time to first occurrence of any of the following clinical events (Composite of any cause death, myocardial infarction, Stroke) within one year follow up.

Secondary variables:

1. Time to the first occurrence of each component of primary clinical events (any cause death, myocardial infarction, Stroke) in the first year after discharge.
2. Proportion of ticagrelor treatment patterns with different clinical outcomes
3. Correlation between risk factors (age, region, education, insurance, hypertension, diabetes, CKD, smoking, etc.) and clinical outcomes

Exploratory variables:

Association between ticagrelor persistence and risk factors (regions, education, reimbursement, etc.); Analysis of other possible factors (such as smoke, LDL-C, etc) affecting the prognosis of patients with ACS; Analysis of possible interactions and their influences between different factors associated with the prognosis of patients with ACS

Exposures of Interest:

Ticagrelor 90 mg used twice a day as part of dual antiplatelet therapy (DAPT) during first year after ACS

Outcomes of Interest:

1. Ticagrelor treatment patterns -Persistence, discontinuation rate, switching and interruption in Chinese ACS patients after hospital discharge;
2. Time of first occurrence of any of the end-point events (any cause death, myocardial infarction, Stroke) within one year follow up.

Limitations:

The study subjects are patients under ticagrelor treatment at discharge in China, which limits the generalization of the study results. The criteria for patients treated with ticagrelor might lead to patient selection bias. As some risk factors of cardiovascular disease (CVD) were not randomized, there might be unmeasured confounding.

ELIGIBILITY:
Inclusion Criteria:

1. ACS patients hospitalized during the following period: from January 2019 to September 2019
2. Patients receiving ticagrelor as part of DAPT at hospital discharge.
3. Patient enrolled into the follow-up program of ACS patients

Exclusion Criteria:

Patients participated in other interventional clinical trials

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ACS patients taking ticagrelor 90 mg twice a day as part of the dual antiplatelet therapy at discharge
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2019-06-19 (Actual); Primary Completion 2021-07-19 (Estimated); Study Completion 2021-07-19 (Estimated)

PRIMARY OUTCOMES:
Ticagrelor persistence | 12 months
  Duration of ticagrelor treatment: Proportion of patients receiving ticagrelor each month after discharge; Duration from the start of treatment to the end of treatment.
Ticagrelor discontinuation and reasons for discontinuation | 12 months
  Percentage of patients with ticagrelor discontinuation and related causes: Discontinuation was defined as stopping P2Y12 for at least 3 months.
Ticagrelor switch and reasons for switching | 12 months
  Percentage of patients with ticagrelor change and related causes: Switching refers to switching from ticagrelor/clopidogrel to another P2Y12 inhibitor (switching from clopidogrel to ticagrelor is a redressing, if documented)
Ticagrelor interruption and reasons for interruption | 12 months
  Percentage of patients with ticagrelor interruption and related causes: Interruptionn was defined as drug withdrawal for more than 1 day and less than 3 months.
Major Adverse Cardiovascular Events | 12 months
  Time to the first occurence of Any cause death, myocardial infarction, or Stroke

SECONDARY OUTCOMES:
Any cause death | 12 months
  Time to the occurence of Any cause death
Myocardial infarction | 12 months
  Time to the first occurence of Myocardial infarction
Stroke | 12 months
  Time to the first occurence of Stroke

CONTACTS AND LOCATIONS:
Overall Officials: Yong Huo, M.D., Principal Investigator — Peking University First Hospital
Locations (1):
- Division of Cardiology, Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hao Y, Liu J, Liu J, Smith SC Jr, Huo Y, Fonarow GC, Ma C, Ge J, Taubert KA, Morgan L, Guo Y, Zhang Q, Wang W, Zhao D; CCC-ACS Investigators. Rationale and design of the Improving Care for Cardiovascular Disease in China (CCC) project: A national effort to prompt quality enhancement for acute coronary syndrome. Am Heart J. 2016 Sep;179:107-15. doi: 10.1016/j.ahj.2016.06.005. Epub 2016 Jun 18. PMID 27595685
- [Background] Valgimigli M, Bueno H, Byrne RA, Collet JP, Costa F, Jeppsson A, Juni P, Kastrati A, Kolh P, Mauri L, Montalescot G, Neumann FJ, Petricevic M, Roffi M, Steg PG, Windecker S, Zamorano JL, Levine GN; ESC Scientific Document Group; ESC Committee for Practice Guidelines (CPG); ESC National Cardiac Societies. 2017 ESC focused update on dual antiplatelet therapy in coronary artery disease developed in collaboration with EACTS: The Task Force for dual antiplatelet therapy in coronary artery disease of the European Society of Cardiology (ESC) and of the European Association for Cardio-Thoracic Surgery (EACTS). Eur Heart J. 2018 Jan 14;39(3):213-260. doi: 10.1093/eurheartj/ehx419. No abstract available. PMID 28886622
- [Background] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846
- [Background] Sun Y, Li C, Zhang L, Hu D, Zhang X, Yu T, Tao M, Wang DW, Shen X. Poor adherence to P2Y12 antagonists increased cardiovascular risks in Chinese PCI-treated patients. Front Med. 2017 Mar;11(1):53-61. doi: 10.1007/s11684-017-0502-2. Epub 2017 Mar 2. PMID 28213881
- [Background] Yeaw J, Benner JS, Walt JG, Sian S, Smith DB. Comparing adherence and persistence across 6 chronic medication classes. J Manag Care Pharm. 2009 Nov-Dec;15(9):728-40. doi: 10.18553/jmcp.2009.15.9.728. PMID 19954264
- [Background] Cramer JA, Roy A, Burrell A, Fairchild CJ, Fuldeore MJ, Ollendorf DA, Wong PK. Medication compliance and persistence: terminology and definitions. Value Health. 2008 Jan-Feb;11(1):44-7. doi: 10.1111/j.1524-4733.2007.00213.x. PMID 18237359